CLINICAL TRIAL: NCT00711373
Title: Vascularized Composite Allotransplantation of the Hand
Acronym: HandCTA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christina L. Kaufman PhD (Other)
Collaborators: Jewish Hospital and St. Mary's Healthcare (Other); Kleinert, Kutz and Associates (Other); University of Louisville (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Christina L. Kaufman PhD, Exec. Director, Christine M. Kleinert Institute for Hand and Microsurgery
Organization: Christine M. Kleinert Institute for Hand and Microsurgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192.98; DoD-OAR A-14022.5
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Upper Extremity Injuries
Keywords: VCA; composite tissue allotransplantation; amputation; Hand

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Unilateral and Bilateral Amputees (Experimental)
  Interventions: Procedure: Allogeneic hand transplantation

INTERVENTIONS:
Procedure: Allogeneic hand transplantation — Surgical reconstruction of part or all of the hands and/or hands and forearm using tissue from a non-living donor

SUMMARY:
This is a clinical trial of unilateral and bilateral hand transplantation. This will be done by the surgical transfer of a hand from a non-living donor to restore function of non-functioning or amputated hand. Recipients must currently take the same type of drugs as a kidney transplant patient to prevent rejection of the hand.

DETAILED DESCRIPTION:
At the Christine M. Kleinert Institute in Louisville, Kentucky, we are recruiting patients for a research protocol that is underway for Composite Tissue Allotransplantation of the Hand. This study is not for all upper extremity injuries, but it is a possibility for some.

The Hand Surgeons at Kleinert, Kutz and Associates and the Christine M. Kleinert Institute performed the first hand transplant in the United States. This patient is doing very well, and is now almost 15 years post transplant. We have also transplanted seven other recipients, including a bilateral recipient. For more information visit www.handtransplant.com.

While hand transplantation is a viable option for select upper extremity amputees, there are significant risks that must be understood before a patient can decide whether hand transplantation is the right option for him or her. The major risk is the systemic immunosuppression that all current hand transplant recipients must take.

As part of this clinical trial of hand transplanation we are also offering a sub-study sub study to determine if cells isolated from fat tissue can be used to control the immune response against the graft. This population of cells that will be isolated from fat tissue is called the stromal vascular fraction (SVF) and has been used on an experimental basis in patients who have problems with blood vessels in their legs, with patients who have received a bone marrow transplant, and with patients who have Chron's disease. These trials have also been experimental. To date, there have been no cases where the SVF cells isolated from and used in the same patient have been associated with harmful side effects.

In this optional sub-study SVF isolated from the patient's own fat tissue would be injected into the graft at the time of transplant, or at the time of a rejection episode. We hope that these cells will help the hand and the nerves heal, and help control your immune systems response against the donor hand. However, this is an experimental study and we don't know if this will work or not. After your transplant and the injection of the SVF cells you will be followed and treated the same as any other hand transplant recipient in this clinical trial.

This sub-study is optional. Subjects can choose to not participate in this sub-study and still be able to participate in the hand transplant clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Candidates may be male or female patients between the ages of 18 and 65 who are missing all or part of a hand and forearm
* No serious co-existing medical or psycho-social problems
* Must be HIV negative at the time of transplant
* Crossmatch is negative between donor and recipient
* Women who are of child bearing potential must have a negative pregnancy test (urine test is acceptable) within 48 hours of transplant and agree to use reliable contraception for one year following transplant
* Subjects must give written informed consent

Exclusion Criteria:

* Uncontrolled infection or severe concomitant diseases which would exclude the recipient from transplantation
* Alcoholism not currently under control
* Malignancy
* Excessive proximal level of amputation: some presence of proximal muscles is required to motor a functioning hand
* Congenital Abnormalities: co-existent absence/atrophy/agenesis of any tissue may affect post transplant results
* History of amputation of less than six months: subject must be allowed to attempt prosthetic use prior to hand transplantation
* Blindness: blind amputees may be poor candidates because sensory return in the hand may not provide sufficient protective sensation
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1998-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
functioning allograft | Monthly functional analysis for first three months and then on an annual basis for the life of the graft
  Subjects will be monitored in Louisville for three months. After that subject will be monitored for function of the allograft on an annual basis or as clinical course indicates. We are requesting that subjects allow function to be evaluated on an annual basis for the life of the graft.

SECONDARY OUTCOMES:
document and manage complications associated with Composite Tissue allotransplantation | monthly labs for the first year, then bi-monthly for the first five years, or as clincial course indicates
  Transplant recipients will have drug levels drawn weekly and then monthly until target blood levels of immunosuppression are acheived. We will then have blood drawn monthly and then quarterly as time progresses. We are requesting that subjects allow us to follow them for the life of the graft.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Jones, MD, Principal Investigator — Jewish Hospital Transplant Center; Tuna Ozyurekoglu, MD, Principal Investigator — Christine M. Kleinert Institute
Locations (1):
- Kleinert Kutz and Associates/Jewish Hospital and St. Mary's Healthcare, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Please visit the above website for more study information. — http://www.handtransplant.com